CLINICAL TRIAL: NCT06258382
Title: Fontan Circulation and Reproductive Health in a National Swedish Cohort
Status: Recruiting | Type: Observational
Sponsor: Caroline Lilliecreutz (Other Government)
Collaborators: Uppsala University (Other); Umeå University (Other); Lund University (Other); Göteborg University (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Caroline Lilliecreutz, MD. PhD, Associate Professor, Linkoeping University
Organization: Linkoeping University (Other Government)
Other Study IDs: 2023-02526-01
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Fontan Circulation
Keywords: reproductive health; cognitive impairment; grown up heart disease
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Male with Fontan circulation: Different data will be collected along with several questionnaires concerning reproductive health. Approximate 100 individuals will be included-
  Interventions: Other: Questionnaires and functional test
- Female with Fontan circulation: Different data will be collected along with several questionnaires concerning reproductive health. Approximate 100 individuals will be included-
  Interventions: Other: Questionnaires and functional test
- Partner to male with Fontan circulation: Different data will be collected along with several questionnaires concerning reproductive health. Approximate 100 individuals will be included-
  Interventions: Other: Questionnaires and functional test
- Partner to female with Fontan circulation: Different data will be collected along with several questionnaires concerning reproductive health. Approximate 100 individuals will be included-
  Interventions: Other: Questionnaires and functional test
- Male control group: Different data will be collected along with several questionnaires concerning reproductive health . Approximate 100 individuals will be included
  Interventions: Other: Questionnaires and functional test
- Female control group: Different data will be collected along with several questionnaires concerning reproductive health. Approximate 100 individuals will be included
  Interventions: Other: Questionnaires and functional test

INTERVENTIONS:
Other: Questionnaires and functional test — Data will be collected from different sources. Questinnaires, Medical journal, Obstetrical records and functional tests

SUMMARY:
In the Swedish registry for congenital heart defects, SWEDCON, over 230 patients with single-ventricle circulation are registered in the adult section.

Congenital heart defects affect career choices, family planning, and leisure activities. Questions regarding heredity and pregnancy are common.

The impact of Fontan circulation on reproductive health and fertility needs to be illuminated, and additional studies are required from both medical and psychosocial perspectives.Cognitive impairment is common among patients with congenital heart defects but is likely an overlooked cause of long-term illness.

Objective To study a large national population (n=200) of adults with Fontan circulation and their potential partners regarding.

* the prevalence and explanatory factors for sexual dysfunction and infertility in women and men with Fontan circulation (Study A).
* the outcomes of pregnancy, choice of delivery mode, and complications in patients with Fontan circulation (Study B).
* the experiences and perceptions of becoming parents among women (n=20) and men (n=20), as well as elucidate reasoning and family planning among women and men (n=20) who have not become parents (Study C).
* Investigate the prevalence and explanatory factors for (Sub-study D):
* Fatigue
* In-depth cognitive screening to describe specific cognitive functions such as auditory memory, visuospatial memory, attention, cognitive speed, and executive functions.

The aim of this research is to gain more knowledge in an area that has been relatively underexplored, thus improving care for women and men with congenital heart defects.

DETAILED DESCRIPTION:
Every year, approximately 2000 children are born with congenital heart defects in Sweden. In a small percentage of these cases, the heart defects are so severe that they cannot be corrected to resemble or function like a healthy heart. Instead, these highly complex heart defects are operated on to establish "single-ventricle circulation," also known as Fontan circulation or TCPC circulation (total cavopulmonary connection). This means there is only one chamber in circulation, pumping blood into the body's main artery. To facilitate venous blood flow to the lungs for oxygenation and back to the heart chamber, high venous pressure and low resistance in the lung circulation are required.

This type of blood circulation can lead to severe complications later in life, including heart failure, low oxygen saturation, blood clot formation, liver cirrhosis, bleeding, protein-losing enteropathy, arrhythmias, and reduced physical capacity. In the Swedish registry for congenital heart defects, SWEDCON, over 230 patients with single-ventricle circulation are registered in the adult section.

Congenital heart defects affect career choices, family planning, and leisure activities. Questions regarding heredity and pregnancy are common. The severity of different heart defects varies and has varying degrees of impact on patients' daily lives. Pregnancy and childbirth exert significant stress on a woman and her body. Due to the increased metabolic needs of the fetus and the mother, hemodynamics change during a normal pregnancy, with approximately a 40-50% increase in cardiac output and plasma volume. Pregnancy is often well tolerated by women with congenital heart defects, but there might be an increased risk of complications associated with pregnancy and childbirth. Women with complex congenital heart defects have a higher risk of experiencing cardiovascular events during pregnancy compared to women with simpler congenital heart defects. There is also a greater risk of infertility for these women. The modified WHO classifications system (mWHO class I-IV) can be used to assess risk associated with pregnancy and childbirth for women with heart disease, where higher class is associated with increased morbidity and mortality. In Fontan circulation, the risk of complications during pregnancy is considered high if the woman is classified as mWHO III or IV. If a woman experiences complications due to Fontan circulation before pregnancy, she is classified as mWHO IV and will be discouraged from pregnancy due to a very high risk for both maternal and fetal complications. During pregnancy, there is an increased risk of arrhythmias, heart failure symptoms, and thrombosis. Miscarriage risk is high for women with Fontan circulation, and preterm delivery is common, often resulting in low birth weight for gestational age. There is also an increased risk of peripartum bleeding. It is recommended that patients with Fontan circulation have frequent check-ups during pregnancy and in the first weeks after delivery.

Some women with complex congenital heart defects choose not to undergo pregnancy due to their heart condition. Others choose to become pregnant despite being informed about the high risks and advice against pregnancy, which places high demands on the care and follow-up of these patients. How men with Fontan circulation perceive their parental abilities and the possibility of having children is poorly studied, as well as how a partner of a person with complex congenital heart defects thinks and reasons about parenthood.

The impact of Fontan circulation on reproductive health and fertility needs to be illuminated, and additional studies are required from both medical and psychosocial perspectives.

Cognitive impairment is common among patients with congenital heart defects but is likely an overlooked cause of long-term illness. Cognitive function and fatigue significantly affect all aspects of quality of life, including employment opportunities, educational level, and the ability to maintain meaningful social relationships, such as marriage. How this affects reproductive health is not fully understood.

Objective:

To study a large national population (n=200) of adults with Fontan circulation and their potential partners regarding.

* the prevalence and explanatory factors for sexual dysfunction and infertility in women and men with Fontan circulation (Study A).
* the outcomes of pregnancy, choice of delivery mode, and complications in patients with Fontan circulation (Study B).
* the experiences and perceptions of becoming parents among women (n=20) and men (n=20), as well as elucidate reasoning and family planning among women and men (n=20) who have not become parents (Study C).
* Investigate the prevalence and explanatory factors for (Sub-study D):
* Fatigue
* In-depth cognitive screening to describe specific cognitive functions such as auditory memory, visuospatial memory, attention, cognitive speed, and executive functions.

Work Plan The study is a national study involving six national centers: Gothenburg, Linköping, Lund, Stockholm, Umeå and Uppsala. Each participating center includes all patients with Fontan circulation. This involves approximately 200 patients and their potential partners.

In Sweden, there are an estimated 40,000 adults with congenital heart defects. We have a unique national register for congenital heart defects, The Swedish Registry of Congenital Heart Disease (SWEDCON), which started in the 1990s with Grown Up Congenital Heart disease (GUCH) and expanded in 2009 to include pediatric cardiology, heart interventions, and now fetal cardiology in congenital heart defects.

Design: Observational study.

The aim of this research is to gain more knowledge in an area that has been relatively underexplored, thus improving care for women and men with congenital heart defects. It is relatively common for women with congenital heart defects to avoid pregnancy due to their heart condition. In cases of aortic valve and/or pulmonary valve disease, Tetralogy of Fallot, and transposition of the great arteries, up to a third of women reported they did not want to have children because of their heart condition .

Therefore, there is significant patient benefit in conducting research among women and men with congenital heart defects. By gaining more knowledge in a new and relatively unexplored area, care can be improved, enabling these women to give birth if they wish without having to avoid it due to their chronic disabilities. Women with less complex heart disease and better functional status can also benefit from new knowledge and improved care, especially since there is a link between maternal congenital heart defects and lower birth weight in infants.

ELIGIBILITY:
Inclusion Criteria:

* Fontan circulation,
* Age ≥18 years at inclusion,
* Follow-up at specialist clinics,
* Ability to fill in questionnaires in the Swedish language (no other alternative available) or
* Partner of a person with Fontan circulation,
* Age ≥18 years at inclusion
* Ability to fill in questionnaires in the Swedish language (no other alternative available).

or •Age- and gender-matched individuals are recruited via the population registry. They must not have congenital heart disease.

Exclusion criteria: N/A

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 200 patients with fontan circulation and their potential partners. Age and gender matched control groups.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence and explanatory factors for sexual dysfunction and infertility in women and men with Fontan circulation | 3 hours
  Reproductive health questionnaire for Woman/reproductive health questionnaire for Man, and a questionnaire for the potential partner, designed for this study.
  International Index of Erectile Function (IIEF5) Female Sexual Function Index (FSFI) EQ-5D is an instrument to describe and measure health and health-related quality of life.

SECONDARY OUTCOMES:
Obstetric, neonatal and cardiological variables before, during, and after pregnancy | 4 hours
  Cardiological complications during pregnancy, at delivery, first 6 months Pregnancy,Obstetric and Neonatal complications e.g.Gestational diabetes, Pregnancy-induced hypertension, Preeclampsia, Anemia,Thromboembolic event, hepatosis, Chorioamnionitis-other Relevant medication. Gestational week at partus Premature delivery Induction with indication, Delivery method; uncomplicated vaginal delivery, instrumental vaginal delivery, Cesarean section,Bleeding (ml) at partus, Birth trauma Placental retention, Maternal death.
  Admission to neonatal ward, Neonatal complications, Child malformations- Type-, Neonatal death, Birth weight, small for gestational age (SGA), large for gestational age (LGA), average for gestational age (AGA) Apgar
Experiences and perceptions of parenthood | 4 hours
  Thoughts, fears, and hopes,Information and knowledge before and during pregnancy, Follow-ups during pregnancy and their extent, Need for special contact at the clinic for congenital heart defects during pregnancy, Physical and mental well-being during and after childbirth ,Describe experiences and perceptions of parenthood in men Long-term follow-up; additional pregnancy, intervention, hospitalization for heart failure/arrhythmia/FALD/endocarditis/infection/stroke, transplantation, cardiovascular death, non-cardiovascular death after 2.5, 10, and 15 years .
  Control group: As control subjects, 200 age- and gender-matched individuals are recruited via the population registry. They must not have congenital heart disease. They will complete the same questionnaires as the study participants and will be asked questions about health status.
Cognitive function | 4 hours
  Multidimensional Fatigue Inventory (MFI-20) Montreal Cognitive Assessment (MoCA) SDMT - Symbol Digit Modalities Test. . TMT A and B - Trail Making Test. BVMT-R - Brief Visuospatial Memory Test. CWIT - Color Word Interference Test. M. FAS - Verbal Fluency Test. DEX - Dysexecutive Questionnaire. . HADs- Hospital Anxiety and Depression Scale BDI II- Beck Depression Inventory

CONTACTS AND LOCATIONS:
Locations (12):
- Sweden (12):
  - Lund University Skåne University Hospital, Lund, Skåne County
  - Sahlgrenska Academy, University of Gothenburg Sahlgrenska University Hospital, Gothenburg
  - Sahlgrenska University Hospital,, Gothenburg
  - University Hospital, Linköping, Linköping
  - Skåne University Hospital, Lund University, Lund
  - Karolinska University Hospital, Stockholm
  - University West, Drottning Silvia's Children's Hospital/Sahlgrenska University Hospital,, Trollhättan
  - Umeå University, Norrland University Hospital, Umeå
  - Umeå University, Norrlands University Hospital, Umeå
  - Akademiska Hospital Uppsala.Uppsala University., Uppsala
  - Uppsala University, Akademiska Hospital, Uppsala
  - Linköping University, University Hospital, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: Undecided